CLINICAL TRIAL: NCT03757260
Title: The Efficacy of Adjunctive Antimicrobial Photodynamic Therapy for Residual Pockets in Previously Surgically Treated Teeth: a Randomized Clinical Trial.
Brief Title: Efficacy of Adjunctive Antimicrobial Photodynamic Therapy for Residual Pockets in Previously Surgically Treated Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Javier Cabrales, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2018:012
Record Dates: First submitted 2018-11-23; First posted 2018-11-28 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Once selected the patient will see two clinicians: the examiner (hygienist) and operator (resident).
  The examiner records the data (PPD, CAL, BOP, PI) of the teeth, and provides preliminary hygiene treatment; the operator delivers the test treatments.
  The treatment assignments are concealed to the patient and the examiner. The operator is unaware of previously recorded data except for pocket depth measurements and is not involved in the post-treatment evaluations (3,6,12 months)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Antimicrobial photodynamic therapy with methylene blue applied to test site after mechanical debridement.
  Interventions: Device: Antimicrobial photodynamic therapy
- Placebo Group (Placebo Comparator): Photodynamic therapy laser is not activated with saline water in the test site after mechanical debridement.
  Interventions: Device: Placebo of photodynamic therapy

INTERVENTIONS:
Device: Antimicrobial photodynamic therapy — Antimicrobial photodynamic therapy is carried out in the residual pockets using the Periowave system. The photosensitizing agent is methylene blue. Approximately 0.2 mL of the solution is applied over 60 seconds to each pocket with a blunt-ended side-port irrigator. The site is illuminated for 60 seconds to activate the agent using a disposable, light-diffusing tip that is introduced into the pocket via a diode laser (wavelength = 675 nm, 160 mW of output power).
  Other Names: "Periowave" trade name
  Arms: Treatment Group
Device: Placebo of photodynamic therapy — The placebo of the antimicrobial photodynamic therapy is carried out in the residual pockets using the Periowave system. The photosensitizing agent is saline solution. Approximately 0.2 mL of the solution is applied over 60 seconds to each pocket with a blunt-ended side-port irrigator. The site is not illuminated (falsely activated) for 60 seconds using a disposable, light-diffusing tip that is introduced into the pocket via a diode laser (wavelength = 675 nm, 160 mW of output power).
  Other Names: Placebo of "Periowave" trade name
  Arms: Placebo Group

SUMMARY:
Traditionally, periodontal gum surgery has been used as a method to gain access to inflamed periodontal pockets around teeth. The outcome of these surgeries, however, is not always successful as there can be recurrence of inflammation and disease. The objective of this study is to assess the effectiveness of antimicrobial photodynamic therapy as an adjunct to mechanical debridement of residual periodontal pockets in patients having undergone periodontal surgery. Pocket probing depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP), and plaque index (PI) will be evaluated at all sites as measures of inflammation and disease resolution.

DETAILED DESCRIPTION:
A single-center, randomized, double-blind, longitudinal study will take place over 12 months. Twenty-eight systemically healthy patients (i.e. absence of uncontrolled diabetes mellitus, cancer, HIV, bone metabolic diseases, or disorders that compromise wound healing) enrolled in a supportive periodontal therapy program and patients at the University of Manitoba Graduate Periodontics Clinic, with at least one surgically treated site with a residual pocket probing depth of ≥ 5mm and bleeding upon probing and having signed the informed consent will be accepted into the study. PPD, CAL, BOP, and PI will be evaluated at these sites. A selected participant will have a full mouth periodontal charting completed prior to baseline measurements as part of their maintenance program.

Once selected the patient will see two clinicians: the examiner (hygienist) and operator (resident).

The examiner records the data (PPD, CAL, BOP, PI) of the entire dentition including the selected tooth or teeth, and provides preliminary hygiene treatment; the operator delivers the test treatments.

The treatment assignments are concealed to the patient and the examiner. The operator is unaware of previously recorded data except for pocket depth measurements and is not involved in the post-treatment evaluations (3,6,12 months). At 12 months, a full mouth re-evaluation will be completed by the examiner as part of the patient's maintenance program.

In the first visit, the examiner records the pocket probing depth, clinical attachment level, presence of bleeding on probing, and plaque index at six sites on involved teeth. Thorough scaling and root planing is performed under local anesthesia using periodontal curettes (Gracey, Hu-Friedy, USA) and an ultrasonic device (Piezo, Ultradent, USA). Once complete, the operator takes over. The patients are then randomly assigned to test or control groups by a computer-generated table. The protocol may be: A, the laser is activated during treatments with methylene blue; B, the laser is never activated during treatments with saline solution.

Antimicrobial photodynamic therapy is carried out in the residual pockets using the Periowave system (Ondine Biomedical Inc, Vancouver, Canada). The photosensitizing agent is methylene blue. Approximately 0.2 mL of the solution is applied over 60 seconds to each pocket with a blunt-ended side-port irrigator. The site is illuminated for 60 seconds to activate the agent using a disposable, light-diffusing tip that is introduced into the pocket via a diode laser (wavelength = 675 nm, 160 mW of output power). The control treatment consists of the same procedure, except that the photosensitizer is replaced with saline solution and the light-diffusing tip is kept in the pocket for 60 seconds without activating the laser. The patient is sent home with a home care package and oral hygiene instructions.

The second session is scheduled after 1 week. The operator applies the photosensitizer and activates the laser according to protocol A or B. The examiner maintains the patients on a 3-month hygiene schedule and reassesses the participants 3, 6, and 12 months after the treatment as well as reinforces oral hygiene instruction. Medical history, concomitant medication, and all adverse events are recorded. Clinical parameters are measured the same way as at baseline. All measurements will be calibrated.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Enrolled in a supportive periodontal therapy program and a patient at the University of Manitoba Graduate Periodontics Clinic
* At least one surgically treated periodontal site with a residual pocket probing depth of ≥ 5mm and bleeding upon probing
* Completed informed consent

Exclusion Criteria:

* Patients with uncontrolled diabetes mellitus
* Patients with cancer
* Patients with HIV
* Patients with bone metabolic diseases
* Patients with disorders that compromise wound healing
* Patients undergoing radiation or immunosuppressive therapy
* Pregnancy or lactation
* Have had antibiotics therapy within the last three months
* Confirmed or suspected intolerance to methylene blue
* Any physical limitations or restrictions that might preclude normal oral hygiene procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in bleeding on probing (BOP) | Initial, 3 months, 6 months, 12 months.
  Change in the presence of bleeding upon probing on individual tooth surfaces at 3 months, 6 months, and 12 months compared to the initial measure.

SECONDARY OUTCOMES:
Change in pocket probing depth (PPD) | Initial, 3 months, 6 months, 12 months.
  Change of the distance from the gingival margin to the tip of the periodontal probe at the bottom of the gingival pocket at 3 months, 6 months, and 12 months compared to the initial measure.
Change of clinical attachment level (CAL) | Initial, 3 months, 6 months, 12 months.
  Change of the distance from the cemento-enamel junction to the tip of the periodontal probe at the bottom of the gingival pocket at 3 months, 6 months, and 12 months compared to the initial measure.
Change of plaque index (PI) | Initial, 3 months, 6 months, 12 months.
  Change in the presence of plaque on individual tooth surfaces at 3 months, 6 months, and 12 months compared to the initial measure.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Cholakis, M Dent, Study Director — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be made available in an anonymized (de-identified) form.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After conclusion of the study up until 5 years after completion of the study.

REFERENCES:
- [Background] Van der Weijden GA, Timmerman MF. A systematic review on the clinical efficacy of subgingival debridement in the treatment of chronic periodontitis. J Clin Periodontol. 2002;29 Suppl 3:55-71; discussion 90-1. doi: 10.1034/j.1600-051x.29.s3.3.x. PMID 12787207
- [Background] Greenstein G. Periodontal response to mechanical non-surgical therapy: a review. J Periodontol. 1992 Feb;63(2):118-30. doi: 10.1902/jop.1992.63.2.118. PMID 1552465
- [Background] Caffesse RG, Sweeney PL, Smith BA. Scaling and root planing with and without periodontal flap surgery. J Clin Periodontol. 1986 Mar;13(3):205-10. doi: 10.1111/j.1600-051x.1986.tb01461.x. PMID 3517073
- [Background] Serino G, Rosling B, Ramberg P, Socransky SS, Lindhe J. Initial outcome and long-term effect of surgical and non-surgical treatment of advanced periodontal disease. J Clin Periodontol. 2001 Oct;28(10):910-6. doi: 10.1034/j.1600-051x.2001.028010910.x. PMID 11686808
- [Background] Mombelli A, Schmid B, Rutar A, Lang NP. Persistence patterns of Porphyromonas gingivalis, Prevotella intermedia/nigrescens, and Actinobacillus actinomyetemcomitans after mechanical therapy of periodontal disease. J Periodontol. 2000 Jan;71(1):14-21. doi: 10.1902/jop.2000.71.1.14. PMID 10695934
- [Background] Magnusson I, Lindhe J, Yoneyama T, Liljenberg B. Recolonization of a subgingival microbiota following scaling in deep pockets. J Clin Periodontol. 1984 Mar;11(3):193-207. doi: 10.1111/j.1600-051x.1984.tb01323.x. PMID 6368611
- [Background] Quirynen M, Bollen CM, Vandekerckhove BN, Dekeyser C, Papaioannou W, Eyssen H. Full- vs. partial-mouth disinfection in the treatment of periodontal infections: short-term clinical and microbiological observations. J Dent Res. 1995 Aug;74(8):1459-67. doi: 10.1177/00220345950740080501. PMID 7560400
- [Background] Sbordone L, Ramaglia L, Gulletta E, Iacono V. Recolonization of the subgingival microflora after scaling and root planing in human periodontitis. J Periodontol. 1990 Sep;61(9):579-84. doi: 10.1902/jop.1990.61.9.579. PMID 2213468
- [Background] Adriaens PA, Edwards CA, De Boever JA, Loesche WJ. Ultrastructural observations on bacterial invasion in cementum and radicular dentin of periodontally diseased human teeth. J Periodontol. 1988 Aug;59(8):493-503. doi: 10.1902/jop.1988.59.8.493. PMID 3171862
- [Background] Kocher T, Fanghanel J, Sawaf H, Litz R. Substance loss caused by scaling with different sonic scaler inserts--an in vitro study. J Clin Periodontol. 2001 Jan;28(1):9-15. doi: 10.1034/j.1600-051x.2001.280102.x. PMID 11142673
- [Background] Flemmig TF, Petersilka GJ, Mehl A, Hickel R, Klaiber B. The effect of working parameters on root substance removal using a piezoelectric ultrasonic scaler in vitro. J Clin Periodontol. 1998 Feb;25(2):158-63. doi: 10.1111/j.1600-051x.1998.tb02422.x. PMID 9495615
- [Background] Ritz L, Hefti AF, Rateitschak KH. An in vitro investigation on the loss of root substance in scaling with various instruments. J Clin Periodontol. 1991 Oct;18(9):643-7. doi: 10.1111/j.1600-051x.1991.tb00104.x. PMID 1960232
- [Background] Zappa U, Smith B, Simona C, Graf H, Case D, Kim W. Root substance removal by scaling and root planing. J Periodontol. 1991 Dec;62(12):750-4. doi: 10.1902/jop.1991.62.12.750. PMID 1765938
- [Background] Badersten A, Nilveus R, Egelberg J. Effect of nonsurgical periodontal therapy. I. Moderately advanced periodontitis. J Clin Periodontol. 1981 Feb;8(1):57-72. doi: 10.1111/j.1600-051x.1981.tb02024.x. PMID 6972954
- [Background] Badersten A, Nilveus R, Egelberg J. Effect of nonsurgical periodontal therapy. II. Severely advanced periodontitis. J Clin Periodontol. 1984 Jan;11(1):63-76. doi: 10.1111/j.1600-051x.1984.tb01309.x. PMID 6363463
- [Background] von Troil B, Needleman I, Sanz M. A systematic review of the prevalence of root sensitivity following periodontal therapy. J Clin Periodontol. 2002;29 Suppl 3:173-7; discussion 195-6. doi: 10.1034/j.1600-051x.29.s3.10.x. PMID 12787217
- [Background] Feres M, Figueiredo LC, Soares GM, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015 Feb;67(1):131-86. doi: 10.1111/prd.12075. PMID 25494600
- [Background] Xue D, Zhao Y. Clinical effectiveness of adjunctive antimicrobial photodynamic therapy for residual pockets during supportive periodontal therapy: A systematic review and meta-analysis. Photodiagnosis Photodyn Ther. 2017 Mar;17:127-133. doi: 10.1016/j.pdpdt.2016.11.011. Epub 2016 Nov 22. PMID 27888165
- [Background] Wilson M. Bactericidal effect of laser light and its potential use in the treatment of plaque-related diseases. Int Dent J. 1994 Apr;44(2):181-9. PMID 8063441
- [Background] Soukos NS, Mulholland SE, Socransky SS, Doukas AG. Photodestruction of human dental plaque bacteria: enhancement of the photodynamic effect by photomechanical waves in an oral biofilm model. Lasers Surg Med. 2003;33(3):161-8. doi: 10.1002/lsm.10208. PMID 12949945
- [Background] Bhatti M, MacRobert A, Meghji S, Henderson B, Wilson M. A study of the uptake of toluidine blue O by Porphyromonas gingivalis and the mechanism of lethal photosensitization. Photochem Photobiol. 1998 Sep;68(3):370-6. PMID 9747591
- [Background] Bhatti M, Nair SP, Macrobert AJ, Henderson B, Shepherd P, Cridland J, Wilson M. Identification of photolabile outer membrane proteins of Porphyromonas gingivalis. Curr Microbiol. 2001 Aug;43(2):96-9. doi: 10.1007/s002840010268. PMID 11391471
- [Background] Harris F, Chatfield LK, Phoenix DA. Phenothiazinium based photosensitisers--photodynamic agents with a multiplicity of cellular targets and clinical applications. Curr Drug Targets. 2005 Aug;6(5):615-27. doi: 10.2174/1389450054545962. PMID 16026282
- [Background] Pfitzner A, Sigusch BW, Albrecht V, Glockmann E. Killing of periodontopathogenic bacteria by photodynamic therapy. J Periodontol. 2004 Oct;75(10):1343-9. doi: 10.1902/jop.2004.75.10.1343. PMID 15562911
- [Background] Chan Y, Lai CH. Bactericidal effects of different laser wavelengths on periodontopathic germs in photodynamic therapy. Lasers Med Sci. 2003;18(1):51-5. doi: 10.1007/s10103-002-0243-5. PMID 12627274
- [Background] Qin YL, Luan XL, Bi LJ, Sheng YQ, Zhou CN, Zhang ZG. Comparison of toluidine blue-mediated photodynamic therapy and conventional scaling treatment for periodontitis in rats. J Periodontal Res. 2008 Apr;43(2):162-7. doi: 10.1111/j.1600-0765.2007.01007.x. PMID 18302617
- [Background] Komerik N, Nakanishi H, MacRobert AJ, Henderson B, Speight P, Wilson M. In vivo killing of Porphyromonas gingivalis by toluidine blue-mediated photosensitization in an animal model. Antimicrob Agents Chemother. 2003 Mar;47(3):932-40. doi: 10.1128/AAC.47.3.932-940.2003. PMID 12604524
- [Background] de Almeida JM, Theodoro LH, Bosco AF, Nagata MJ, Oshiiwa M, Garcia VG. Influence of photodynamic therapy on the development of ligature-induced periodontitis in rats. J Periodontol. 2007 Mar;78(3):566-75. doi: 10.1902/jop.2007.060214. PMID 17335382
- [Background] Braun A, Dehn C, Krause F, Jepsen S. Short-term clinical effects of adjunctive antimicrobial photodynamic therapy in periodontal treatment: a randomized clinical trial. J Clin Periodontol. 2008 Oct;35(10):877-84. doi: 10.1111/j.1600-051X.2008.01303.x. Epub 2008 Aug 17. PMID 18713259
- [Background] Christodoulides N, Nikolidakis D, Chondros P, Becker J, Schwarz F, Rossler R, Sculean A. Photodynamic therapy as an adjunct to non-surgical periodontal treatment: a randomized, controlled clinical trial. J Periodontol. 2008 Sep;79(9):1638-44. doi: 10.1902/jop.2008.070652. PMID 18771363
- [Background] Andersen R, Loebel N, Hammond D, Wilson M. Treatment of periodontal disease by photodisinfection compared to scaling and root planing. J Clin Dent. 2007;18(2):34-8. PMID 17508621
- [Background] Chondros P, Nikolidakis D, Christodoulides N, Rossler R, Gutknecht N, Sculean A. Photodynamic therapy as adjunct to non-surgical periodontal treatment in patients on periodontal maintenance: a randomized controlled clinical trial. Lasers Med Sci. 2009 Sep;24(5):681-8. doi: 10.1007/s10103-008-0565-z. Epub 2008 May 9. PMID 18465191
- [Background] Muller Campanile VS, Giannopoulou C, Campanile G, Cancela JA, Mombelli A. Single or repeated antimicrobial photodynamic therapy as adjunct to ultrasonic debridement in residual periodontal pockets: clinical, microbiological, and local biological effects. Lasers Med Sci. 2015 Jan;30(1):27-34. doi: 10.1007/s10103-013-1337-y. Epub 2013 May 10. PMID 23660738
- [Background] Campos GN, Pimentel SP, Ribeiro FV, Casarin RC, Cirano FR, Saraceni CH, Casati MZ. The adjunctive effect of photodynamic therapy for residual pockets in single-rooted teeth: a randomized controlled clinical trial. Lasers Med Sci. 2013 Jan;28(1):317-24. doi: 10.1007/s10103-012-1159-3. Epub 2012 Jul 20. PMID 22814896
- [Background] Cappuyns I, Cionca N, Wick P, Giannopoulou C, Mombelli A. Treatment of residual pockets with photodynamic therapy, diode laser, or deep scaling. A randomized, split-mouth controlled clinical trial. Lasers Med Sci. 2012 Sep;27(5):979-86. doi: 10.1007/s10103-011-1027-6. Epub 2011 Nov 22. PMID 22105837
- [Background] de Paula Eduardo C, de Freitas PM, Esteves-Oliveira M, Aranha AC, Ramalho KM, Simoes A, Bello-Silva MS, Tuner J. Laser phototherapy in the treatment of periodontal disease. A review. Lasers Med Sci. 2010 Nov;25(6):781-92. doi: 10.1007/s10103-010-0812-y. Epub 2010 Jul 17. PMID 20640471
- [Background] Jori G, Fabris C, Soncin M, Ferro S, Coppellotti O, Dei D, Fantetti L, Chiti G, Roncucci G. Photodynamic therapy in the treatment of microbial infections: basic principles and perspective applications. Lasers Surg Med. 2006 Jun;38(5):468-81. doi: 10.1002/lsm.20361. PMID 16788934